CLINICAL TRIAL: NCT02443571
Title: A Retrospective Observational Study Investigating the Safety and Effectiveness of Fluciclovine (18F) (FACBC) PET Ligand in Human Subjects
Brief Title: Retrospective Observational Study Investigating Fluciclovine (18F) (FACBC)
Status: Completed | Type: Observational
Sponsor: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: Fluciclovine (18F) - BED - 001
Record Dates: First submitted 2015-05-11; First posted 2015-05-14 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Prostatic Neoplasms
Keywords: observational study
MeSH Terms: conditions — Prostatic Neoplasms | interventions — fluciclovine F-18

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Fluciclovine (18F) — Not applicable. This is an observational study.
  Other Names: FACBC

SUMMARY:
This retrospective observational multi centered study has been established to collect the clinical experience relating to the administration of Fluciclovine 18F employed in both investigator initiated studies and named patient/compassionate use programmes in up to 5 sites.

DETAILED DESCRIPTION:
This study will collect clinical data from consenting patients (unless a HIPAA waiver or equivalent was granted) who received the PET radiotracer Fluciclovine 18F (FACBC) (a synthetic amino acid analog) for imaging of patients with various cancers at participating sites in the US and Europe.

Data collection will cover baseline medical history and medications in all patients.

The result of PET radiotracer and other imaging findings, and reports of histopathology from biopsied tissue (where available) and in a time window relevant to the use of PET imaging in the diagnosis of primary/recurrent prostate cancer will be recorded.

In all subjects, with regards to safety monitoring, available data for physical examination, vital signs and laboratory test results will be collected from 28 days prior to and out to a 35 day window after Fluciclovine 18F (FACBC) administration.

The major goals of the investigation are to consolidate the safety profile of Fluciclovine 18F (FACBC), to evaluate its use in the detection of local and extraprostatic recurrence of prostate cancer and to evaluate its ability to detect malignancy in patients undergoing screening for primary prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient managed by a site at which ethical committee approval for retrospective data collection under this protocol has been received
* Patient has received at least one injection of fluciclovine (18F) for the detection of a malignant tumour at any location

Exclusion Criteria:

* Subjects will be excluded from the analyses if any of the following criteria are met:
* Patients participating in clinical trials or open access programmes at countries or sites not participating in this study.
* Patients managed at sites without ethical committee approval for retrospective data collection under this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients (male/female) who underwent PET scanning using fluciclovine (18F) as the radiotracer for the detection of cancer at a clinical site participating in this study.
Sampling Method: Non-Probability Sample
Enrollment: 714 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Penelope Ward, MBBS FFPM, Study Chair — Blue Earth Diagnostics
Locations (4):
- Emory University Hospital, Atlanta, Georgia, United States
- University Hospital Sant'Orsola Malpighi, Bologna, Italy
- Norway (2):
  - Oslo University Hospital, Oslo
  - Aleris Kreftsenter, Oslo

REFERENCES:
- [Result] Bach-Gansmo T, Nanni C, Nieh PT, Zanoni L, Bogsrud TV, Sletten H, Korsan KA, Kieboom J, Tade FI, Odewole O, Chau A, Ward P, Goodman MM, Fanti S, Schuster DM, Willoch F. Multisite Experience of the Safety, Detection Rate and Diagnostic Performance of Fluciclovine (18F) Positron Emission Tomography/Computerized Tomography Imaging in the Staging of Biochemically Recurrent Prostate Cancer. J Urol. 2017 Mar;197(3 Pt 1):676-683. doi: 10.1016/j.juro.2016.09.117. Epub 2016 Oct 13. PMID 27746282

RESULTS

PARTICIPANT FLOW:
Groups:
- Recurrent Prostate Cancer: Recurrent Prostate Cancer
- Primary Prostate Cancer: Primary Prostate Cancer
- Other Cancers: Other Cancers
Period: Overall Study
Arm/Group | Recurrent Prostate Cancer | Primary Prostate Cancer | Other Cancers
Started | 596 | 95 | 23
Completed | 596 | 95 | 23
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Recurrent Prostate Cancer | Primary Prostate Cancer | Other Cancers | Total
Number analyzed (Participants) | 596 | 95 | 23 | 714
Age, Continuous [Mean (Full Range); unit: Years] | 67 [42 to 90] | 65 [44 to 88] | 61 [34 to 89] | 66 [34 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 16 | 16
  Male | 596 | 95 | 7 | 698
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 26 | 0 | 3 | 29
  White | 186 | 0 | 17 | 203
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 382 | 95 | 3 | 480
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 137 | 10 | 21 | 168
  Norway | 371 | 85 | 2 | 458
  Italy | 88 | 0 | 0 | 88

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events and Treatment-Emergent Serious Adverse Events
Description: Treatment-emergent Adverse Events and Treatment-Emergent Serious Adverse Events
Time Frame: Up to 35 days post Fluciclovine 18F
Population: Patients who have received at least one dose of Fluciclovine 18F
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrent Prostate Cancer | Primary Prostate Cancer | Other Cancers
Number analyzed (Participants) | 596 | 95 | 23
Participants
  Treatment Emergent Adverse Events | 32 | 2 | 8
  Treatment Emergent Serious Adverse Events | 1 | 1 | 0

2. Primary Outcome: Positive Predictive Value of FACBC Compared to Histology to Detect Recurrence in Patients Previously Diagnosed With Prostate Cancer
Description: Positive Predictive Value is the percentage of participants with a positive Fluciclovine 18F scan who truly have positive finding in biopsy.
Time Frame: Up to 1 year post Fluciclovine 18F
Population: Standard of truth was histology. For the prostate/bed region standard TRUS/biopsy or MRI/TRUS fusion biopsy was used to establish truth while blinded to PET findings.
  When feasible, clinically relevant 18F-fluciclovine positive extraprostatic areas underwent directed biopsy based on cognitive fusion of the PET/CT data with biopsy technique.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Recurrent Prostate Cancer
Number analyzed (Participants) | 143
Percentage of participants
  Subject PPV | 82.4 [74.3 to 88.7]
  Extraprostatic Region PPV: number analyzed (Participants) | 44
  Extraprostatic Region PPV | 92.3 [79.1 to 98.4]
  Prostate & Prostate Bed Region PPV: number analyzed (Participants) | 127
  Prostate & Prostate Bed Region PPV | 71.8 [62.1 to 80.3]

3. Primary Outcome: Positive Predictive Value of FACBC to Detect Presence of Malignant Disease in Patients Undergoing Screening for Primary Prostate Cancer
Description: as for outcome 2
Time Frame: Up to 1 year post Fluciclovine 18F
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Primary Prostate Cancer
Number analyzed (Participants) | 61
Percentage of participants | 100 [93.7 to 100]

4. Secondary Outcome: Detection Rate, Sensitivity, Specificity, and Negative Predictive Value in Biochemically Recurrent Prostate Cancer
Description: Detection rate is the percentage of participants with positive finding in Fluciclovine 18F scan.
  Sensitivity is the percentage of participants with positive finding in biopsy correctly identified as positive by Fluciclovine 18F scan.
  Specificity is the percentage of participants with negative finding in biopsy correctly identified as negative by Fluciclovine 18F scan.
  Negative Predictive Value is the percentage of participants with a negative Fluciclovine 18F scan who truly don't have positive finding in biopsy.
Time Frame: Up to 1 year post Fluciclovine 18F
Measure: Number (95% Confidence Interval); unit: Percentages
Arm/Group | Recurrent Prostate Cancer
Number analyzed (Participants) | 125
Percentages
  Detection Rate | 82.4 [74.6 to 88.6]
  Sensitivity | 94.7 [88.0 to 98.3]
  Specificity | 54.8 [36.0 to 72.7]
  Negative Predictive Value | 77.3 [54.6 to 92.2]

5. Secondary Outcome: Detection Rate, Sensitivity, Specificity, and Negative Predictive Value to Detect Presence of Malignant Disease in Patients Undergoing Screening for Primary Prostate Cancer
Description: as for outcome 4
Time Frame: Up to 1 year post Fluciclovine 18F
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Primary Prostate Cancer
Number analyzed (Participants) | 61
Percentage of participants
  Detection Rate | 93.4 [84.1 to 98.2]
  Sensitivity | 93.4 [84.1 to 98.2]

ADVERSE EVENTS:
Time Frame: All Treatment Emergent Adverse Events (TEAEs) occurring up to 35 days after each 18F-fluciclovine administration, and for all TEAEs occurring between two consecutive administrations of 18F and up to 35 days after the last 18F administration.
Groups:
- 18F-Fluciclovine PET: 18F-Fluciclovine PET
Arm/Group | 18F-Fluciclovine PET
All-Cause Mortality (participants affected / at risk) | 0/714
Serious Adverse Events (participants affected / at risk) | 2/714
Other Adverse Events (participants affected / at risk) | 9/714
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 18F-Fluciclovine PET (N=714)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1
Post Procedural Pulmonary Embolism (Injury, poisoning and procedural complications) | 1
Hypertension (Vascular disorders) | 1
Blood Pressure Decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 18F-Fluciclovine PET (N=714)
Injection site extravasation (General disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No